CLINICAL TRIAL: NCT01246622
Title: Phase I Trial of Cytarabine and Lenalidomide in Relapsed or Refractory Acute Myeloid Leukemia Patients
Brief Title: Lenalidomide and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 179510; NCI-2010-02080 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-11-12; First posted 2010-11-23 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Cytarabine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (biological therapy) (Experimental): Patients receive lenalidomide PO on days 6-26 and cytarabine IV over 3 hours on days 1-5. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cytarabine; Drug: lenalidomide

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid

SUMMARY:
This phase I trial is studying the side effects and best dose of lenalidomide when given together with cytarabine in treating patients with relapsed or refractory acute myeloid leukemia (AML). Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with cytarabine may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of lenalidomide following intermediate dose ARA-C (cytarabine) in relapsed/refractory AML.

SECONDARY OBJECTIVES:

I. Evaluate immune reconstitution in patients in complete remission (CR) treated at the MTD.

II. Evaluate the efficacy of the regimen in the expanded group treated at the MTD.

OUTLINE: This is a dose-escalation study of lenalidomide.

Patients receive lenalidomide orally (PO) on days 6-26 and cytarabine intravenously (IV) over 3 hours on days 1-5. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed/refractory AML for which no standard effective therapy is anticipated to result in a durable partial or complete remission
* Eastern Cooperative Oncology Group Performance (ECOG) status 0-2
* Bilirubin =< 2.5 x upper limit of normal (ULN) unless considered Gilbert's syndrome of leukemia
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN unless considered Gilbert's syndrome of leukemia
* Partial thromboplastin time (PTT) must be < 1.5 x ULN and international normalized ratio (INR) < 1.5 ULN
* Phase I subjects must have calculated creatinine clearance >= 50 ml/min by Cockcroft-Gault formula
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by RevAssist) of lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Patient is capable of understanding and complying with parameters as outlined in the protocol and able to sign informed consent
* For patients with thromboembolic risk (history of deep venous thrombosis [DVT]/pulmonary embolism [PE], on medications that increase risk of thrombolic event, etc.) able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin [ASA] may use warfarin or low molecular weight heparin); the risk of blood clots may also be increased when lenalidomide is combined with other drugs known to cause blood clots such as steroids, other forms of cancer drugs, hormone replacement therapy, birth control pills and erythropoietin

Exclusion Criteria:

* Known active central nervous system (CNS) disease
* The patient has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic or any investigational agents within 14 days or 5 half lives, whichever is greater, prior to drug administration on this study or has not recovered to less than grade 2 clinically significant non-hematological adverse effects/toxicities of the previous therapy except hydroxyurea up to 24 hours prior to cytarabine initiation
* The patient has a documented left ventricular ejection fraction of < 50 %
* Active uncontrolled infection
* Symptomatic congestive heart failure
* Unstable angina pectoris or cardiac arrhythmia
* History of adrenal insufficiency
* Psychiatric illness/social situation that would limit compliance with study requirements
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are seropositive because of hepatitis B virus vaccine are eligible
* Any medical condition which in the opinion of the study investigator places the patient at an unacceptable high risk of toxicities
* Lactating or pregnant female (Lactating females must agree not to breast feed while taking lenalidomide)
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments or any other investigational agent except hydroxyurea up to 24 hours prior to cytarabine initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02-07 (Actual); Primary Completion 2014-05-15 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide following intermediate dose cytarabine | Over course 1
  Assessed by Cancer Therapy Evaluation Program (CTEP) Version 4 of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Overall response rate | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Griffiths, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States